CLINICAL TRIAL: NCT00782639
Title: RECARE (REnal Safety Following the Intra-Arterial Administration of Iopamidol vs. Iodixanol During Coronary AngiogRaphy in DiabEtic Patients)
Brief Title: Renal Safety of Iopamidol Versus Iodixanol During Coronary Angiography in Diabetic Patients
Acronym: RECARE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated early due to slow enrollment.
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP114
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Results first posted 2011-09-01 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Renal Impairment; Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Iopamidol; iodixanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iopamiro-370 (Active Comparator)
  Interventions: Drug: Iopamidol injection 76%
- Visipaque 320 (Active Comparator)
  Interventions: Drug: iodixanol

INTERVENTIONS:
Drug: Iopamidol injection 76% — Iopamiro-370 (Iopamidol injection 76%) is provided in single dose bottles/vials, ready to use, aqueous, nonpyrogenic, colorless to pale yellow sterile solution
  Other Names: Isovue
  Arms: Iopamiro-370
Drug: iodixanol — Visipaque 320 (iodixanol) injection is provided in bottles/flexible containers, ready to use sterile, pyrogen-free colorless to pale yellow solution
  Arms: Visipaque 320

SUMMARY:
The purpose of this study is to compare the incidence of contrast-induced nephropathy (CIN) following the administration of iopamidol-370 (Iopamiro-370) and iodixanol-320 (Visipaque 320) in patients with moderate-to-severe chronic kidney disease and diabetes mellitus undergoing cardiac angiography.

DETAILED DESCRIPTION:
This was a Phase IV, multicenter, randomized, double-blind, parallel-group comparison of iopamidol-370 and iodixanol-320 in patients at high risk for CIN, i.e., patients with:

* Stage 3 or 4 CKD (SCr level of ≥ 1.5 mg/dL for men and ≥1.3 mg/dL for women or eGFR between 15 and 50 mL/min, and
* Diabetes mellitus who would undergo clinically indicated cardiac angiography procedures. Approximately 10 investigative centers were to participate in this study. This study was to enroll approximately 220 patients to ensure that 200 evaluable patients were able to complete the study according to this protocol.

Patients were to be randomized to receive either iopamidol-370 or iodixanol-320. Each patient was to be evaluated for the occurrence of CIN within 48 to 72 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Provides written Informed Consent and is willing to comply with protocol requirements
* Is >18 years of age
* Has a documented predose serum creatinine level of ≥1.5 mg/dL for men and ≥1.3 mg/dL for women or predose eGFR of >15 and ≤50 mL/min/1.73 m2, calculated via the Modification of Diet in Renal Disease (MDRD) formula from a SCr obtained within 72 hours of enrollment into the study;
* Diagnosed as having diabetes mellitus (Type 1 or Type 2) treated with insulin or oral hypoglycemic agents for at least 6 months
* Is referred for cardiac angiography with or without percutaneous coronary intervention;
* If at the discretion of the Investigator is receiving or will be receiving a prophylactic medication for renal function, the medication is one that is permitted by this protocol (N acetylcysteine, 1200 mg twice daily on the day before and on the day of the cardiac angiography procedure);
* Undergoes or is scheduled to undergo pre, peri, or post procedure hydration permitted by this protocol, i.e.:

  154 mEq/L sodium bicarbonate solution, administered intravenously at 3 mL/kg/hr for 1 hour before cardiac angiography, followed by an infusion of 1 mL/kg/hr during and out to 6 hours after cardiac angiography, or 154 mEq/L sodium chloride solution (0.9% normal saline), administered intravenously at 1 mL/kg/hr for 8 12 hours before cardiac angiography, followed by an infusion of 1 mL/kg/hr during and out to 8-12 hours after cardiac angiography

Exclusion Criteria:

-Is a pregnant or lactating female. Exclude the possibility of pregnancy: by laboratory testing on-site at the institution (measurement of serum or urine beta human chorionic gonadotropin) within 24 hours prior to the start of investigational product administration by history (e.g., tubal ligation or hysterectomy, post menopausal with a minimum 1 year without menses)

* Has a history of hypersensitivity to iodine-containing compounds;
* Has unstable renal function (i.e., acute worsening of renal function, as determined by the Investigator, that has been observed in the 7 days prior to enrollment) and/or is in acute renal failure;
* Has stage 5 chronic kidney disease or end-stage renal disease (i.e., estimated glomerular filtration rate [eGFR] <15 mL/min/1.73 m2)
* Has severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association (NYHA);
* Has uncontrolled diabetes, as determined by the Investigator;
* Has received an iodinated contrast agent within 7 days prior to the administration of the study agent or is scheduled to receive an iodinated contrast agent within 72 hours after administration of the study agent;
* Is receiving cyclo-oxygenase-2 inhibitors, nonsteroidal anti-inflammatory drugs (with exception of low dose aspirin [≤325 mg per day]), aminoglycosides, or any other drugs that carry a significant risk of nephrotoxicity (in the opinion of the Investigator) during the time period beginning within 72 hours prior to contrast administration and up to 72 hours postdose;
* Prior to, during or post the cardiac angiography, is receiving or will be receiving a prophylactic medication to prevent acute kidney injury that is not permitted by this protocol (e.g., theophylline, fenoldopam, etc.);
* During cardiac angiography, is going to receive provocative pharmacological agents such as adenosine or dipyridamole;
* Is planned to undergo major surgery (e.g. coronary artery bypass graft, valve surgery, etc.) within 48-72 hours after contrast administration;
* Is planned to receive an intravenous diuretic or mannitol as prophylaxis to prevent acute renal injury (Note: chronic administration is allowed);
* Is hemodynamically unstable within 48 hours pre-contrast administration defined as a systolic blood pressure <90 mmHg or requires pressor or intra-aortic balloon support;
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or postdose follow-up examinations;
* Is determined by the Investigator that the patient is clinically unsuitable for the study Note: Changes in diuretics, angiotensin-converting enzyme inhibitors, or angiotensin receptor blockers doses within 72 hours prior to and up to 72 hours post contrast administration should be avoided unless clinically necessary for the subject's underlying medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Spinazzi, M.D., Study Chair — Bracco Diagnostics
Locations (1):
- Bracco Diagnostics Inc., Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 4 investigational centers in China. The first subject was enrolled on 24 March 2009, and the last subject completed the study on 06 September 2009.
Pre-assignment Details: Phase IV, multicenter, randomized, double-blind, parallel-group comparison of iopamidol-370 and iodixanol-320 in patients at high risk for CIN (patients with Stage 3 or 4 CKD [men: SCr level of ≥1.5 mg/dL; women: ≥1.3 mg/dL or eGFR between 15 and 50 mL/min]) & Diabetes mellitus who would undergo clinically indicated cardiac angiography procedures.
Groups:
- Iopamiro-370: (Iopamidol injection at the 370 mgI/mL concentration)
- Visipaque 320: (Iodixanol injection at the 320 mgI/mL concentration)
Period: Overall Study
Arm/Group | Iopamiro-370 | Visipaque 320
Started | 12 | 11
Completed | 12 (This study was terminated due to low enrollment.) | 11 (This study was terminated due to low enrollment.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iopamiro-370 | Visipaque 320 | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  China | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Contrast-induced Nephropathy (CIN)
Description: The number of participants who presented with CIN (defined as an increase in Serum Creatinine (SCr) from baseline greater than or equal to 0.5 mg/dL following the administration of iopamidol-370 or iodixanol 320 while undergoing cardiac angiography). Since CIN is a prospectively-defined outcome measure of the trial, patients experiencing CIN were not reported as having an adverse event.
Time Frame: 48 to 72 hours After Injection of Contrast Media
Measure: Number; unit: Participants
Arm/Group | Iopamiro-370 | Visipaque 320
Number analyzed (Participants) | 12 | 11
Participants | 1 | 0

2. Secondary Outcome: The Number of Participants With a >=25% Decrease in Estimated Glomerular Filtration Rate (eGFR)
Description: This outcome measure provides the total number of participants that had a decrease from baseline in eGFR greater or equal to 25% within 48 to 72 hours following the cardiac angiography procedure.
Time Frame: Baseline (just prior to injection of contrast media) and 48 to 72 hours after injection of contrast media
Measure: Number; unit: Participants
Arm/Group | Iopamiro-370 | Visipaque 320
Number analyzed (Participants) | 12 | 11
Participants | 1 | 0

3. Secondary Outcome: The Number of Participants With a >=25% Increase in Serum Creatinine (SCr)
Description: This outcome measure provides the total number of participants that had a increase from baseline in SCr greater or equal to 25% within 48 to 72 hours following the cardiac angiography procedure.
Time Frame: Baseline (just prior to injection of contrast media) and 48 to 72 hours after injection of contrast media
Measure: Number; unit: Participants
Arm/Group | Iopamiro-370 | Visipaque 320
Number analyzed (Participants) | 12 | 11
Participants | 1 | 0

4. Secondary Outcome: Number of Participants Requiring Dialysis
Description: This outcome measure provides the total number of participants requiring dialysis occurring from acute renal failure.
Time Frame: 48 to 72 hours after injection of contrast media
Measure: Number; unit: Participants
Arm/Group | Iopamiro-370 | Visipaque 320
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Who Died From Acute Renal Failure
Description: This outcome measure provides the total number of participants who died as a result of acute renal failure.
Time Frame: Any timepoint (Screening [up to 72 hours prior to injection of contrast media], Baseline [just before injection], or 48 to 72 hours or 7 days after injection)
Measure: Number; unit: Participants
Arm/Group | Iopamiro-370 | Visipaque 320
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

6. Primary Outcome: Baseline and Change From Baseline Measurements for the One Participant With Contrast-Induced Nephropathy (CIN) at the 48 to 72 Hours After Injection of Contrast Media Visit
Description: Only 1 participant presented with incidence of CIN (change from baseline greater than or equal to 0.5 mg/dL) following the administration of iopamidol-370 while undergoing cardiac angiography. The participant's measurements at baseline and at 48 to 72 hours after the injection of contrast agent, as well as the difference between the two, are displayed here. Since CIN is a prospectively-defined outcome measure of the trial, patients experiencing CIN were not reported as having an adverse event.
Time Frame: Baseline (just prior to injection of contrast media) and 48 to 72 hours after injection of contrast media
Measure: Number; unit: milligrams per deciliter (mg/dL)
Groups:
- Iopamiro-370: (Iopamidol injection at the 370 milligrams of iodine per milliliter [mgI/mL] concentration)
- Visipaque 320: (Iodixanol injection at the 320 milligrams of iodine per milliliter [mgI/mL] concentration)
Arm/Group | Iopamiro-370 | Visipaque 320
Number analyzed (Participants) | 1 | 0
milligrams per deciliter (mg/dL)
  Baseline | 1.10 |
  48 to 72 hours After Injection of Contrast Media | 1.60 |
  Change from Baseline | 0.50 |

ADVERSE EVENTS:
Time Frame: Subjects were monitored for any untoward medical occurrences ("adverse events") from the time of signed informed consent and enrollment into the study ("Screening") through 2 hours after the last injection of contrast media.
Description: As CIN was a prospectively-defined outcome measure of the trial, patients experiencing CIN were not reported as having an adverse event.
Arm/Group | Iopamiro-370 | Visipaque 320
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
This study was terminated early due to low enrollment. Only 1 patient in the Iopamiro-370 group had CIN (per all 3 definitions [first 3 secondary outcome measures] of CIN); therefore, no formal analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be presented during scientific symposia or published in a scientific journal only after review by Bracco in accordance with the guidelines set forth in the applicable publication or financial agreement.